CLINICAL TRIAL: NCT05779735
Title: Validation of Ultrasound "Angle of Progression" Measurement to Decrease the Cesarean Rate : a Randomized Comparative Multicenter Prospective Study.
Brief Title: Validation of Ultrasound "Angle of Progression" Measurement to Decrease the Cesarean Rate
Acronym: DELIVERY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A01978-35 DELIVERY
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Prolonged Second Stage of Labor
Keywords: angle of progression; cesarean delivery; transperineal ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : control (No Intervention): The mode of delivery will be determined by clinical examens (digital examination)
- Group 2 : Transperineal ultrasound measurements of AOP (Experimental): The mode of delivery will be determined by clinical examens (digital examination) and ultrasound measurement of the AOP :
  * vaginal delivery is encouraged if AOP measurement is >120°
  * cesarean delivery is encouraged if AOP measurement is <= 120°
  Interventions: Diagnostic Test: Transperineal ultrasound measurements of AOP

INTERVENTIONS:
Diagnostic Test: Transperineal ultrasound measurements of AOP — The angle of progression (AOP) defined as the angle between the pubic bone axis and the leading part of the fetal head
  Arms: Group 2 : Transperineal ultrasound measurements of AOP

SUMMARY:
Ultrasound during labor and measurement of Angle of progression showed extensive prospective and retrospective publications since 2010. The investigators performed between 2013 and 2016 the only one multicenter, randomized controlled Trial comparing digital exam to angle of progression after a prolonged 2-hour second stage of labor with uncertain fetal head. The investigators consider a cut off of 120° to accepted vaginal birth among cephalic occiput anterior position This randomised PILOT study showed that measurement of Angle of progression in addition to digital exam reduced caesarean delivery from 41% to12% ( n= 33, p=0,06). doi: 10.1016/j.ajog.2022.04.018.

The objective of this new study is therefore to validate the results of this PILOT study in a more powerful multicenter randomized trial (DELIVERY).

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous or multiparous women with no history of vaginal delivery,
* > or = 37 weeks amenorrhoea
* Cephalic presentation in anterior position (occipito-pubic position, left anterior occipito-iliac and right anterior occipito-iliac ) confirmed by ultrasound
* uncertain fetal head engagement on digital examination or midline fetal presentation in prolonged second stage of labor (at least 2 hours),

Exclusion Criteria:

* Multiparous women who were previous vaginal deliveries,
* Presentation other than cephalic,
* Twin pregnancies,
* Posterior or transverse position
* Transperineal ultrasound for head-perineum distance measurement
* Fetal heart rate abnormalities requiring rapid delivery,
* Contraindication to vaginal delivery whether maternal or fetal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-09-13 (Estimated); Study Completion 2025-10-13 (Estimated)

PRIMARY OUTCOMES:
cesarean delivery rate | baseline
  Demonstrate that the angle of progression measurement would change by 20% the cesarean rate after a prolonged second stage of labor (2 hours).

SECONDARY OUTCOMES:
Number of complicated deliveries in each group | baseline
  A complicated deliveries is defined by the occurrence of at least one of the following events :
  * Failed instrumental extraction
  * Sequential use of a second instrument,
  * Difficult instrumental extraction defined as :
    * vacuum detachment
    * requires the use of a second instrument,
    * extraction time > 10 minutes,
    * operator's impression of the difficulty of extraction,
  * Shoulder dystocia by obstetric maneuver
Severe maternal morbidity, in each group | 1 month
  Severe maternal morbidity is defined by the occurrence of at least one of the following events:
  * postpartum hemorrhage requiring hysterectomy, embolization, conservative surgical treatment or blood transfusion,
  * third or fourth degree perineal tears
  * vaginal thrombus,
  * cervical tear,
  * surgical wounds
  * sepsis, amniotic embolism, cardiac complication or renal failure.
Severe neonatal morbidity, in each group | 1 month
  Severe neonatal morbidity, in each group, defined by the occurrence of at least one event below:
  * severe biological signs
  * moderate or absent biological signs but associated with perinatal events
  * seizure
  * severe neonatal trauma
  * Fetal death or neonatal death.
Rate of admission to neonatal intensive care unit, in each group | 1 month
  Number of newborns admitted to intensive care out of the total number of newborns
Concordance rate between the routinely AOP measurement and the centralized AOP measurement reading | 1 month
  Centralized blind AOP measurement reading

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Haumonte, Principal Investigator — Hopital Saint Joseph Marseille
Locations (7):
- France (7):
  - CHU de Lille - Hôpital Jeanne de Flandre, Lille
  - APHM Hôpital Conception, Marseille
  - Hopital Saint Joseph, Marseille
  - APHM Hôpital Nord, Marseille
  - Hôpital Armand Trousseau AP-HP, Paris
  - CHIC Poissy, Poissy
  - CHITS Hôpital Sainte Musse, Toulon